CLINICAL TRIAL: NCT03561103
Title: Impact of Representative Payee Services on ART Adherence Among Marginalized People Living With HIV/AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Mary Hawk, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY20110364; 1R01MH112416-01A1 (NIH)
Record Dates: First submitted 2018-05-22; First posted 2018-06-19 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: The study includes an RCT with two randomized arms plus additional non-randomized arms.
  In the RCT, 160 participants will be recruited. The RCT consists of an Intervention group that receives client-centered representative payee services in addition to standard of care; the control group receives standard of care only.
  For the two additional non-randomized ("Choice") arms, two arms have been added through which an additional 50 people will be recruited. The Choice Intervention arm (n=25) receives client-centered representative payee services in addition to standard of care. The Choice control group (n=25) receives standard of care. Participant in the choice arms are not randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RCT: Intervention (Experimental): Participants in the RCT intervention arm will receive client-centered representative payee services in addition to the standard of care.
  Interventions: Behavioral: Client-Centered Representative Payee
- RCT: Control (No Intervention): Participants in the RCT control group will receive the standard of care.
- Choice Intervention (Experimental): Participants in the Choice intervention arm will receive client-centered representative payee services in addition to the standard of care. They will not be randomly assigned.
  Interventions: Behavioral: Client-Centered Representative Payee
- Choice Control (No Intervention): Participants in the RCT control group will receive the standard of care. They will not be randomly assigned.

INTERVENTIONS:
Behavioral: Client-Centered Representative Payee — CCRP is a structural intervention wherein Social Security authorizes a representative payee to serve as financial manager for people who need help managing their money. By helping clients to consistently pay their bills including rents and utilities, CCRP may redirect the expenditure of participants' resources toward improved health behaviors. Shifting the focus of material and biopsychosocial resources may change the context in which health behaviors are produced, contributing to higher rates of adherence and viral suppression. CCRP modifies the implementation of a current policy of the Social Security Administration (SSA) to create an intervention that is highly replicable.
  Arms: Choice Intervention; RCT: Intervention

SUMMARY:
Client-Centered Representative Payee is a structural intervention that provides financial management support to PLWHA by modifying the implementation of a long-standing policy within the Social Security Administration, in which an organization is authorized to serve as the client's payee. The central hypothesis of this study is that by helping clients to pay rent and other bills on time, housing stability will improve and financial stress will decrease. By reducing the cognitive burden of living with chronic financial stress and frequent threats of housing loss, clients can devote more time and attention to medical appointments and medication adherence. It is further hypothesized that these changes will improve clients' self-efficacy for health behaviors, retention in care, medication adherence, and viral loads. These hypotheses will be tested via the following specific aims: (1) Conduct a randomized controlled trial with two randomized arms (n=160) and two non-randomized arms (n=50) to test the effect of Client-Centered Rep Payee on ART adherence and viral load among PLWHA who are economically disadvantaged and unstably housed. Clinical adherence will be compared through behavioral and biological measures including prescription refill data, self-reported appointment adherence, and viral load for patients receiving the intervention versus those receiving standard of care. (2) Test underlying mechanisms associated with Client-Centered Rep Payee that contribute to changes in medication adherence and viral suppression rates. This will be accomplished via use of quantitative (mediation analysis) and qualitative (semi-structured interview) methods to test hypothesized mediators of medication adherence and viral suppression including financial and housing instability, financial stress, self-efficacy for health behaviors, and retention in care. (3) Assess the cost and cost-effectiveness of the Client-Centered Rep Payee model. An economic analysis will be conducted to model the impact of the intervention as compared with standard of care on quality adjusted life years as well as new infections averted. This approach is innovative because it offers a structural intervention to improve adherence by addressing the effects of economic insecurity, requires low financial investment, and can be layered with existing clinical services. Further, it is highly scalable as it builds on a current policy in practice within the Social Security system.

DETAILED DESCRIPTION:
Marginalized populations, including those who are unstably housed and have mental health or substance use disorders, demonstrate alarming rates of disparities in the incidence of new HIV infections and treatment outcomes. These populations have HIV viral suppression rates as low as 13% and mortality 3 to 5 times higher than people living with HIV/AIDS (PLWHA) who have stable housing. Economic disadvantage can contribute to poor medication adherence and clinical outcomes through limited social resources, repeated cycles of housing instability, high levels of stress caused by financial insecurity, and lack of resources to cope with these demands. While the remediation of poverty on a broad scale is not on the near horizon, addressing factors that result from economic disadvantage and limit adherence is feasible and achievable. The investigators aim to understand whether providing financial management to marginalized PLWHA can improve their financial and housing stability, and in turn, antiretroviral therapy treatment adherence and rates of viral suppression.

Representative payee is a structural intervention that provides financial management to marginalized individuals, which has already shown promise in helping marginalized populations achieve undetectable viral loads. Structural interventions aim to alter social, political, or economic contexts in order to improve health outcomes rather than focusing on proximal health behaviors (14). "rep payee" is a Social Security Administration (SSA) policy whereby an organization is appointed to serve as a money manager for vulnerable individuals who receive SSA benefits. The client and their physician complete a request for determination of a representative payee, and once authorized bu SSA, the rep payee establishes a checking account for the client into which SSA entitlements are directly deposited. The client does not have direct access to the account. The rep payee pays the client's bills, which improves regular payment of rent and utilities, and then disburses expendable funds to the client.

In a pilot study examining associations between our "Client-Centered rep payee" services and viral load, it was found that only 7 of 18 participants had suppressed viral loads (SVL) at baseline, but 16 of the 18 had SVL at six-month follow-up (p = .004, McNemar's) (15). In a more recent analysis, investigators determined that of 40 participants who received Client Centered rep payee, 82% had suppressed viral loads at both 6- and 12-months follow up. The Open Door, Inc. (TOD), the organization that developed this intervention, has provided these services to 76 PLWHA over the past nine years. Though clients can terminate the rep payee arrangement at any time, 90% of clients has kept TOD as their rep payee indefinitely, demonstrating both the feasibility and acceptability of this approach. The hypothesis is that by helping clients to pay their rent and other bills on time, housing stability improves and financial stress decreases. By reducing the cognitive burden of living with chronic financial stress and frequent threats of housing loss, clients can devote more time and attention to medical appointments and medication adherence. Ultimately, it is believed that this program improves clients' self-efficacy for health behaviors, retention in care, medication adherence, CD4 counts, and viral loads. These these hypotheses will be tested via the following aims in a randomized controlled trial of 320 PLWHA.

Aim 1. Conduct a randomized controlled trial (RCT, n=160) with two additional non-randomized arms (n=50) to test the effect of Client-Centered Rep Payee on anti-retroviral (ART) medication adherence and viral load among PLWHA who are economically disadvantaged and unstably housed. Compare clinical adherence will be assessed through behavioral and biological measures including, self-reported appointment adherence, and viral load for patients receiving the intervention versus those receiving standard of care.

Aim 2. Test underlying mechanisms associated with Client-Centered Rep Payee that contribute to changes in medication adherence and viral suppression rates. Quantitative (mediation analysis) and qualitative (semi-structured interview) methods will be used to test hypothesized mediators of medication adherence and viral suppression including financial and housing instability, financial stress, self-efficacy for health behaviors, and retention in care.

Aim 3. Assess the cost and cost-effectiveness of the Client-Centered Rep Payee model. The investigators will conduct an economic analysis to model the impact of the intervention as compared with standard of care on quality adjusted life years as well as new infections averted.

Client-Centered Rep Payee offers a structural intervention to improve adherence by addressing economic insecurity. This approach requires low financial investment and can be layered with existing clinical services. Further, it is highly scalable as it builds on a current policy in practice within the Social Security system. It is projected that by demonstrating the impact and cost-effectiveness of Client-Centered Rep Payee an innovative approach to improving viral suppression rates and reducing health disparities among marginalized PLWHA may be documented.

ELIGIBILITY:
Inclusion Criteria:

* Living with HIV/AIDS
* 18 years of age and older
* English- or Spanish-speaking
* Recipient of Social Security entitlements (SSI and/or SSDI)
* Income below 138% of the federal poverty level
* One or more of the following: Not virally suppressed (viral suppression is denoted at 200 copies/ml); Unsustained viral suppression over the past 12 months; Poor ART adherence. Poor ART adherence is assessed via a CASE Index Score ≤10 or via a single question to assess the percentages of missed doses in the past week <90%. (New clients who do not have historical viral load data but are not suppressed at baseline will be eligible for the study if they meet other criteria.)
* Able and willing to provide informed consent

Exclusion Criteria:

* Currently receiving Representative Payee services or having received them in the past 12 months.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Change in ART Adherence | Baseline, 12-months
  Change in ART adherence will be calculated by comparing HIV viral load counts at Baseline versus 12 months.

SECONDARY OUTCOMES:
Persistence of change in ART Adherence | Baseline plus 12 months versus Baseline plus 24 months.
  Persistence of change in ART adherence will be calculated by comparing HIV viral load counts at 12 versus 24 months.
ART Adherence | Self-report of ART adherence will be measured at Baseline, 6-, and 12-months.
  Self-report of ART adherence will be measured via the CASE adherence index, which captures self-reported missed doses of medicine.
CD4 | CD4 will be collected at Baseline, 6-, 12-, 18-, and 24- months.
  CD4 counts will be used to assess immune system functioning.
Self-efficacy for Adherence | Self-efficacy for adherence will be measured at Baseline, 6-, and 12-months.
  Self-efficacy for adherence assess the participants' perception that they can take their medications as prescribed even in times of duress. This will be measured via HIV-ASES, (Johnson, 2007), a 12-item scale designed to assess self-efficacy for taking HIV medications
Retention in Care | Retention in Care will be measured at Baseline, 6-, and 12-months.
  Retention in Care assess the number of missed versus total scheduled visits. Retention is defined by having at least one primary care visit per quarter or two kept visits separated by ≥ 90 days.
Health-Related Quality of Life | Health-Related Quality of Life will be measured at Baseline, 6-, and 12-months.
  Quality of Life related to health will be measured by a single Item General Health Measure (SF-12; DiSalvo, 2006), which is, "In general, would you say your health is: (Excellent, Very good, Good, Fair, Poor)."
Self-report of Financial Stress | Self-report of financial stress will be measured at Baseline, 6-, and 12-months.
  This measure assesses the participant's self-report of stress related to financial challenges such as late payments, growing debt, etc. It will be assessed via the Financial measures from Background Stress Inventory (Terrill, 2015).
Social Support | Social support will be measured at Baseline, 6-, and 12-months.
  Emotional, informational and tangible functional forms of social support will be measured via the Medical Outcomes Study Social Support Survey (MOS-SSS).
Housing Status I | Housing status I will be measured at Baseline, 6-, and 12-months.
  Participants' self-reported housing status will be measured via a single item question "Which best describes your current living situation?" (Stably Housed/Unstably House/Homeless) as found in Wolitski, et. al., 2010.
Housing Status II | Housing Status II will be measured at Baseline, 6-, and 12-months.
  A second measure of housing status, newly developed by the study team, will be assessed via the following two questions: "In the past 90 days, have you (1) Received an eviction notice or notice to vacate because your rent was not paid? (2) Had your utilities shutoff because your bill was not paid?"
Experiences of Payeeship | Experiences of Payeeship will be measured at Baseline, 6-, and 12-months.
  A 17-item questionnaire with 4 subscales will be used to assess participants (a) Satisfaction with payee/case manager, (b) Involvement of beneficiary in money management, (c) Perceived benefit from payee arrangement, and (d) feeling coerced. These questions have been modified from a previous study (Rosen et. al., 2005).
Substance Use | Substance use behaviors will be measured at Baseline, 6-, and 12-months.
  Changes in substance use behaviors will be measured via the Risk Assessment Battery (Metzger, et.a., 1993).
Sexual Risk | Sexual Risk will be assessed at Baseline, 6-, and 12-months.
  Sexual risk behaviors will be assessed to determine the likelihood of infecting others with HIV. This will be measured via the Risk Assessment Battery (Metzger, et.a., 1993).
Depressive Symptoms | Depressive Symptoms will be measured at Baseline, 6-, and 12-months.
  Individuals experience of depressive symptoms will be measured via the Quick Inventory of Depressive Symptomology (Rush, et.al., 2003).
Connections with Providers | Connections with Providers will be measured at Baseline, 6-, and 12-months.
  The Health Care Relationship Trust Scale will be used to assess the patient-provider relationship; i.e., discussion options, committed to best care, interested in me as a person, excellent listener, accepts me, tells me complete truth, trusts me as an individual, makes me feel I am worthy of his/her time, takes time to listen, comfort talking about personal issues, feel better after seeing healthcare provider (Bova, 2012).

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Hawk, DrPH, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - Birmingham AIDS Outreach, Birmingham, Alabama
  - Action Wellness, Philadelphia, Pennsylvania
  - The Open Door, Inc., Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olaniyan A, Creasy SL, Batey DS, Brooks MM, Maulsby C, Musgrove K, Hagan E, Martin D, Sashin C, Farmartino C, Hawk M. Protocol of a randomized controlled trial to test the effects of client-centered Representative Payee Services on antiretroviral therapy adherence among marginalized people living with HIV. BMC Public Health. 2020 Sep 23;20(1):1443. doi: 10.1186/s12889-020-09500-z. PMID 32967646

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/03/NCT03561103/Prot_SAP_004.pdf